CLINICAL TRIAL: NCT03391609
Title: Peri-operative Dexmedetomidine Infusion in Mild Pre-eclamptic Patients Undergoing Elective Cesarean Section Under General Anesthesia
Brief Title: Peri-operative Dexmedetomidine Infusion in Pre-eclamptic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, lecturer, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 144
Record Dates: First submitted 2017-12-18; First posted 2018-01-05 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control group (Placebo Comparator): Caesarian section will be performed under standard general anesthesia plus pre and intra operative saline infusion (placebo) in the same rate as dexmedetomedine starting 15 minutes before induction of general anesthesia and continue till peritoneum closure.
  Interventions: Drug: placebo infusion
- Dex. group (Active Comparator): Caesarian section will be performed under standard general anesthesia plus pre and intra operative Dexmedetomidine infusion in a dose of 0.5mic/kg/hour starting 15 minutes before induction of general anesthesia and continue till peritoneum closure.
  Interventions: Drug: Dexmedetomidine infusion

INTERVENTIONS:
Drug: placebo infusion — Caesarian section will be performed under standard general anesthesia plus pre and intra operative saline infusion (placebo) in the same rate as dexmedetomedine starting 15 minutes before induction of general anesthesia and continue till peritoneum closure.
  Arms: control group
Drug: Dexmedetomidine infusion — Caesarian section will be performed under standard general anesthesia plus pre and intra operative Dexmedetomidine infusion in a dose of 0.5mic/kg/hour starting 15 minutes before induction of general anesthesia and continue till peritoneum closure.
  Arms: Dex. group

SUMMARY:
The purpose of this study is to investigate the effects of dexmedetomidine infusion on the stress response to intubation, postoperative analgesia, and renal functions (urinary output [UOP], creatinine and glomerular filtration rate [GFR]) in preeclamptic patient.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* have mild preeclampsia ( Pre-eclamptic patients will be defined as having hypertension [systolic blood pressure (SBP) ≥140 mmHg and/or diastolic blood pressure (DBP)≥90 mmHg] accompanied by proteinuria first detected after 20 weeks of gestation).
* Proteinuria is defined as at least 300 mg protein in 24 h urine collection [or ≥1+ dipstick (30 mg/dl) in a single urine sample] ).
* American Society of Anesthesiologists (ASA) physical status of II or III.
* age between 19 and 40 years

Exclusion Criteria:

* patient refusal to consent (obsolete).
* pre-existing neurological disease or psychic patients.
* history of cardiac and respiratory system failure.
* co-existing significant renal or liver disease.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-18 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
postoperative analgesia | 24 hours postoperatively
  through VAS score readings

SECONDARY OUTCOMES:
stress response | 24 hours postoperatively
  mean arterial blood pressure
renal function | 24 hours postoperatively
  glomerular filtration rate
untoward events | 24 hours postoperatively
  eclampsia, drug side effects (over sedation, hypotension, bradycardia)

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt